CLINICAL TRIAL: NCT04341376
Title: Embedding Mental Health Consultation Within Prenatal Home Visiting to Prevent Child Maltreatment and Violence Exposure
Brief Title: Prevention of Childhood Maltreatment in Families With Young Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CE003103 (NIH)
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Child Maltreatment; Child Exposure to Intimate Partner Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced First Connections (Experimental): Enhanced First Connections is a short-term risk assessment and response home visiting referral program. The goal of Enhanced First Connections is to identify family needs and link families to community resources, including evidence based home visiting models. Enhanced First Connections includes prenatal identification and engagement of women with an adversity or trauma history, and infant and early childhood mental health consultation. Women who enroll in Enhanced First Connections are expected to receive between four and eight home visits before being referred to other community resources.
  Interventions: Behavioral: Enhanced First Connections
- Treatment as Usual (No Intervention): Women who receive Treatment as Usual will follow the usual course of clinical care throughout their pregnancy and into the postpartum period, and will be eligible for the typical array of community services that may be offered to them.

INTERVENTIONS:
Behavioral: Enhanced First Connections — Enhanced First Connections is a short-term home visiting program that includes prenatal identification and engagement of women with an adversity or trauma history, and infant and early childhood mental health consultation.
  Arms: Enhanced First Connections

SUMMARY:
This study will examine the efficacy of Enhanced First Connections, which is a short-term perinatal home visiting program that includes infant and early childhood mental health consultation. Mothers with a history of adversity or trauma will be the focus of this research. Hypothesized outcomes of Enhanced First Connections include the prevention of child maltreatment (child abuse and neglect), prevention of child exposure to adult intimate partner violence, increases in family engagement in longer-term evidence based home visiting programs, increases in family engagement in specialized support services to address maternal adversity and trauma, reductions in maternal risk factors, and the promotion of positive parenting and the parent-child relationship.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Recruited in the second or third trimester of pregnancy
* At least one self-reported experience of adversity or trauma
* English or Spanish speaking

Exclusion Criteria:

- Does not meet all inclusion criteria above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 200 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Child Maltreatment Status | 6-months postpartum
  Child protection record review
Child Exposure to Intimate Partner Violence | 6-months postpartum
  Child protection record review
Maternal Report of Intimate Partner Violence | 6-months postpartum
  Maternal report: Conflict Tactics Scales

SECONDARY OUTCOMES:
Family engagement in evidence based home visiting programs | 6-months postpartum
  Home visiting record review
Contextual stress exposure | 6-months postpartum
  Maternal report: Contextual Stress Interview
Maternal depressive symptoms | 6-months postpartum
  Maternal report: Patient Health Questionnaire-9
Maternal anxiety symptoms | 6-months postpartum
  Maternal report: Generalized Anxiety Disorder 7-item scale
Maternal PTSD symptoms | 6-months postpartum
  Maternal report: Short Post-Traumatic Stress Disorder Rating Interview
Maternal alcohol use | 6-months postpartum
  Maternal report: Alcohol Use Disorders Test
Maternal substance use | 6-months postpartum
  Maternal report: Drug Abuse Screening Test
Maternal parenting stress | 6-months postpartum
  Maternal report: Parenting Stress Index
Maternal sensitivity | 6-months postpartum
  Observation of free play interaction coded using Parent Caregiver Involvement Scales and Emotional Availability Scales
Maternal hostility | 6-months postpartum
  Observation of free play interaction coded using Emotional Availability Scales
Maternal non-responsiveness | 6-months postpartum
  Maternal report: Maternal Responsiveness Questionnaire
Home environment | 6-months postpartum
  Home Observation for Measurement of the Environment
Mother-infant relationship | 6-months postpartum
  Maternal report: Postpartum Bonding Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie H Parade, PhD, Principal Investigator — E.P. Bradley Hospital
Locations (1):
- E.P. Bradley Hospital, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets generated from questionnaire, interview, and observational assessments will be cleaned and merged using SPSS syntax to generate a final dataset for analysis. A public use de-identified dataset that does not include sensitive or potentially identifiable information will be made available. For datasets that include sensitive or potentially identifiable information, data-use agreements will be put in place with appropriate restrictions prior to the provision of data. To ensure that released data have appropriate documentation, a data dictionary will accompany all de-identified datasets that includes data collection methods, measures and variable construction, and potential limitations of use.
Supporting Information: Study Protocol, SAP
Time Frame: A de-identified dataset will be made available within 30 months following completion of the project or at the time of the publication of manuscripts that present the main aims of the study
Access Criteria: A public use de-identified dataset that does not include sensitive or potentially identifiable information will be made broadly available. For datasets that include sensitive or potentially identifiable information, data-use agreements will be put in place with appropriate restrictions prior to the provision of data.